CLINICAL TRIAL: NCT04711109
Title: BRCA-P: A Randomized, Double-Blind, Placebo-Controlled, Multi-Center, International Phase 3 Study to Determine the Preventive Effect of Denosumab on Breast Cancer in Women Carrying a BRCA1 Germline Mutation
Brief Title: Studying the Effect of Denosumab on Preventing Breast Cancer in Women With a BRCA1 Germline Mutation
Acronym: BRCA-P
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Austrian Breast & Colorectal Cancer Study Group (ABCSG) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: A211801; NCI-2020-11358 (Registry Identifier: NCI Clinical Trial Reporting Program); UG1CA189823 (NIH); 2017-002505-35 (EudraCT Number); ABCSG 50 (Other: Austrian Breast & Colorectal Cancer Study Group)
Record Dates: First submitted 2021-01-13; First posted 2021-01-15 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: BRCA1 Mutation; Breast Cancer; Breast Diseases; Breast Neoplasms; Breast Carcinoma; Neoplasms
Keywords: RANKL; Breast Cancer Prevention; Denosumab; Bone Density Conservation Agents; Physiological Effects of Drugs
MeSH Terms: conditions — Breast Neoplasms; Breast Diseases; Neoplasms | interventions — Denosumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A (denosumab) (Experimental): Patients receive denosumab SC q6m for up to 5 years in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Denosumab; Other: Quality-of-Life Assessment
- Arm B (placebo) (Placebo Comparator): Patients receive placebo SC q6m for up to 5 years in the absence of disease progression.
  Interventions: Drug: Placebo; Other: Quality-of-Life Assessment

INTERVENTIONS:
Drug: Denosumab — Given SC
  Arms: Arm A (denosumab)
Drug: Placebo — Given SC
  Arms: Arm B (placebo)
Other: Quality-of-Life Assessment — Ancillary studies

SUMMARY:
This phase III trial compares denosumab to placebo for the prevention of breast cancer in women with a BRCA1 germline mutation. A germline mutation is an inherited gene change which, in the BRCA1 gene, is associated with an increased risk of breast and other cancers. Denosumab is a monoclonal antibody that is used to treat bone loss in order to reduce the risk of bone fractures in healthy people, and to reduce new bone growths in cancer patients whose cancer has spread to their bones. Research has shown that denosumab may also reduce the risk of developing breast cancer in women carrying a BRCA1 germline mutation.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the reduction in the risk of any breast cancer (invasive or ductal carcinoma in situ [DCIS]) in women with germline BRCA1 mutation who are treated with denosumab compared to placebo.

SECONDARY OBJECTIVES:

I. To determine the reduction in the risk of invasive breast cancer in women with germline BRCA1 mutation who are treated with denosumab compared to placebo.

II. To determine the reduction in the risk of invasive triple negative breast cancer (TNBC) in women with germline BRCA1 mutation who are treated with denosumab compared to placebo.

III. To determine the reduction in risk of ovarian, fallopian and peritoneal cancers (in women who have not undergone prophylactic bilateral salpingo-oophorectomy [PBSO]) in women with germline BRCA1 mutation who are treated with denosumab compared to placebo.

IV. To determine the reduction in risk of other (i.e. non-breast and nonovarian) malignancies, including those known to be associated with BRCA1 germline mutations in women with germline BRCA1 mutation who are treated with denosumab compared to placebo.

V. To determine the reduction in the risk of clinical fractures in pre- and postmenopausal women with germline BRCA1 mutation who are treated with denosumab compared to placebo.

VI. To compare rates of breast biopsies and rate of benign breast lesions in women with germline BRCA1 mutation who are treated with denosumab compared to placebo.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM A: Patients receive denosumab subcutaneously (SC) every 6 months (q6m) for up to 5 years in the absence of the development of breast cancer or unacceptable toxicity.

ARM B: Patients receive placebo SC q6m for up to 5 years in the absence of the development of breast cancer.

After completion of study treatment, patients are followed up every 12 months for 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Women with a confirmed deleterious or likely deleterious BRCA 1 germline mutation (variant class 4 or 5)
* Age >= 25 years and =< 55 years at randomization
* No evidence of breast cancer by MRI or mammography (MG) and clinical breast examination within the last 6 months prior to randomization
* No clinical evidence of ovarian cancer at randomization
* Negative pregnancy test at randomization for women of childbearing potential
* No preventive breast surgery planned at time of randomization
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Written informed consent before any study-specific procedure is performed

Exclusion Criteria:

* Prior bilateral mastectomy
* History of ovarian cancer (including fallopian and peritoneal cancer)
* History of breast cancer
* History of invasive cancer except for basal cell or squamous cell skin cancer or carcinoma in situ of the cervix, stage 1 papillary or follicular thyroid cancer, atypical hyperplasia or LCIS (lobular carcinoma in situ)
* Pregnant or lactating women (within the last 2 months prior to randomization)
* Unwillingness to use highly effective contraception method during and within at least 5 months after cessation of denosumab/placebo therapy in women of childbearing potential. (Note: Women of childbearing potential should be monitored for pregnancy prior to each denosumab/placebo injection)
* Clinically relevant hypocalcemia (history and current condition), or serum calcium < 2.0 mmol/L (< 8.0 mg/dL)

  * Hypocalcemia defined by calcium below the normal range (a single value below the normal range does not necessarily constitute hypocalcemia, but should be 'corrected' before dosing the subject). Monitoring of calcium level in regular intervals (usually prior to investigational product [IP] administration) is highly recommended
* Tamoxifen, raloxifene or aromatase inhibitor use during the last 3 months prior to randomization or for a duration of more than 3 years in total (current and prior hormone replacement therapy [HRT] is permitted)
* Prior use of denosumab
* Subject has a known prior history or current evidence of osteonecrosis or osteomyelitis of the jaw, or an active dental/jaw condition which requires oral surgery including tooth extraction within 3 months of enrollment
* Concurrent treatment with a bisphosphonate or an anti-angiogenic agent
* Any major medical or psychiatric condition that may prevent the subject from completing the study
* Known active infection with hepatitis B virus or hepatitis C virus
* Known infection with human immunodeficiency virus (HIV)
* Use of any other investigational product (current or prior aspirin or non-steroidal anti-inflammatory drugs [NSAIDs] are permitted)

Ages: 25 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 300 (Estimated)
Dates: Start 2023-02-14 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2033-12 (Estimated)

PRIMARY OUTCOMES:
Time to the occurrence of any breast cancer (invasive or ductal carcinoma in situ [DCIS]) | From randomization to the occurrence of breast cancer (invasive or DCIS), assessed up to 5 years
  Time to breast cancer (invasive or DCIS) will be compared between the two treatment arms using a stratified Cox proportional hazards regression model.

SECONDARY OUTCOMES:
Time to invasive breast cancer | Up to 5 years post treatment
  Will be compared between the two treatment arms using a stratified Cox proportional hazards regression model.
Time to invasive triple negative breast cancer | Up to 5 years post treatment
  Will be compared between the two treatment arms using a stratified Cox proportional hazards regression model.
Time to ovarian, fallopian and peritoneal cancer (in women who have not undergone prophylactic bilateral salpingo-oophorectomy) | Up to 5 years post treatment
  Will be compared between the two treatment arms using a stratified Cox proportional hazards regression model. Time to ovarian cancer will be analyzed in the overall group and in different strata (oral contraceptive use, hormone replacement therapy use, and menopausal status).
Time to other (nonbreast or ovarian cancer) malignancies, including those known to be associated with BRCA1 mutations | Up to 5 years post treatment
  Will be compared between the two treatment arms using a stratified Cox proportional hazards regression model.
Time to clinical fractures in pre- and postmenopausal women | Up to 5 years post treatment
  Will be compared between the two treatment arms using a stratified Cox proportional hazards regression model.
Frequency of breast biopsies | Up to 5 years post treatment
  May be recommended as part of care based on a finding on mammogram, MRI, ultrasound or physical exam performed as part of monitoring for breast cancer. Will be compared between the two treatment arms via chi-square analysis.
Frequency of benign breast lesions | Up to 5 years post treatment
  May be recommended as part of care based on a finding on mammogram, MRI, ultrasound or physical exam performed as part of monitoring for breast cancer. Will be compared between the two treatment arms via chi-square analysis.
Assess incidence, nature and severity of adverse events (AEs) using the National Cancer Institute Common Terminology Criteria for Adverse Events version 4.0 | Up to 5 years post treatment
  Overall toxicity rates (percentages) for grade 3 or higher adverse events considered at least possibly related to treatment will be reported per treatment arm.

CONTACTS AND LOCATIONS:
Overall Officials: Judy E. Garber, MD, MPH, Study Chair — Dana-Farber Cancer Institute
Locations (47):
- United States (47):
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - UCSF Medical Center-Mount Zion, San Francisco, California
  - Rocky Mountain Cancer Centers-Aurora, Aurora, Colorado
  - UCHealth University of Colorado Hospital, Aurora, Colorado
  - Rocky Mountain Cancer Centers-Boulder, Boulder, Colorado
  - Rocky Mountain Cancer Centers - Centennial, Centennial, Colorado
  - Rocky Mountain Cancer Centers-Midtown, Denver, Colorado
  - Rocky Mountain Cancer Centers-Rose, Denver, Colorado
  - Mountain Blue Cancer Care Center - Swedish, Englewood, Colorado
  - Rocky Mountain Cancer Centers - Swedish, Englewood, Colorado
  - Rocky Mountain Cancer Centers-Littleton, Littleton, Colorado
  - Rocky Mountain Cancer Centers-Sky Ridge, Lone Tree, Colorado
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - Northwestern University, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - NorthShore University HealthSystem-Evanston Hospital, Evanston, Illinois
  - NorthShore University HealthSystem-Highland Park Hospital, Highland Park, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - University of Kansas Hospital-Indian Creek Campus, Overland Park, Kansas
  - University of Kansas Hospital-Westwood Cancer Center, Westwood, Kansas
  - Maine Medical Center- Scarborough Campus, Scarborough, Maine
  - Maine Medical Partners - South Portland, South Portland, Maine
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Corewell Health Grand Rapids Hospitals - Butterworth Hospital, Grand Rapids, Michigan
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - OptumCare Cancer Care at Fort Apache, Las Vegas, Nevada
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Novant Health Presbyterian Medical Center, Charlotte, North Carolina
  - Novant Health Breast Surgery - Greensboro, Greensboro, North Carolina
  - Novant Health Cancer Institute - Kernersville, Kernersville, North Carolina
  - Novant Health Cancer Institute - Mount Airy, Mount Airy, North Carolina
  - Novant Health Cancer Institute - Thomasville, Thomasville, North Carolina
  - Novant Health Forsyth Medical Center, Winston-Salem, North Carolina
  - Sanford Roger Maris Cancer Center, Fargo, North Dakota
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - University of Pennsylvania/Abramson Cancer Center, Philadelphia, Pennsylvania
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - University of Vermont Medical Center, Burlington, Vermont
  - Virginia Commonwealth University/Massey Cancer Center, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: Yes